CLINICAL TRIAL: NCT03482154
Title: Malglycemia in the Pediatric Hematopoietic Stem Cell Transplant Population
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 16-1496.cc
Record Dates: First submitted 2018-03-15; First posted 2018-03-29 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Stem Cell Transplant Complications; Hyperglycemia; Hypoglycemia
MeSH Terms: conditions — Hyperglycemia; Hypoglycemia | interventions — Stem Cell Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With Malglycemia
  Interventions: Procedure: Hematopoietic Stem Cell Transplant
- Without Malglycemia
  Interventions: Procedure: Hematopoietic Stem Cell Transplant

INTERVENTIONS:
Procedure: Hematopoietic Stem Cell Transplant — Allogeneic and autologous stem cell transplants covering both malignant and non-malignant diagnoses.

SUMMARY:
This is a retrospective chart review of patients who underwent a hematopoietic stem cell transplant (HSCT) between 1994 and 2016 to evaluate incidence of malglycemia and the relationship to specific outcomes.

DETAILED DESCRIPTION:
This is a retrospective chart review of patients who underwent a hematopoietic stem cell transplant between 2007 and 2016 to evaluate incidence and risk factors of malglycemia. The review will also aim to characterize relationships between specific outcomes and malglycemia in pediatric HSCT patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 0 to 30 years old at time of transplant
* Bone Marrow Transplant (BMT) recipient at Children's Hospital Colorado (CHCO) between 1/1/2007 and 7/31/2016

Exclusion Criteria:

* Preexisting diabetes mellitus or known hyperglycemia
* Inadequate blood glucose data for analysis

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients who received hematopoietic stem cell transplants with the Bone Marrow Transplant Program at Children's Hospital Colorado from January 1, 2007 to July 31, 2016.
Sampling Method: Non-Probability Sample
Enrollment: 344 (Actual)
Dates: Start 2016-09-06 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patients experiencing malglycemia in primary admission for pediatric HSCT patients | Transplant Day -14 to +100
  hypoglycemia (BG < 70 mg/dL), hyperglycemia (BG ≥ 126 mg/dL), or glycemic variability (σ ≥ 29 mg/dL)
Number of patients with versus without malglycemia who experience infection | Transplant Day 0 to +100
  It is hypothesized that patients who experience malglycemia will have an increased rate of post-transplant infections. This outcome will be assessed for differences in incidence based on malglycemia occurence

SECONDARY OUTCOMES:
Determine whether specific exposures are associated with increased occurrence of malglycemia | Transplant Day -14 to +100
  The occurrence of the outcome, malglycemia, with be assessed for differences in incidence that may occur as a result of age, medication exposures (use of glucocorticoids, asparaginase, total parenteral nutrition (TPN), or calcineurin inhibitors), underlying diagnosis, and transplant type
Survival rate of patients with versus without malglycemia | Transplant Day 0 through date of relapse or death
  It is hypothesized that patients who experience malglycemia will have an increased rate of post-transplant mortality. This outcome will be assessed for differences in incidence based on malglycemia occurrence
Occurrence of graft-versus-host disease (GVHD) in patients with versus without malglycemia | Transplant Day 0 through date of relapse or death
  It is hypothesized that patients who experience malglycemia will have an increased rate of GVHD. This outcome will be assessed for differences in incidence based on malglycemia occurrence

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Sopfe, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho S, Vigers T, Pyle L, Franklin A, Sopfe J, Jeney F, Forlenza G. Composite Metric of Glycemic Control Q-Score Is Elevated in Pediatric and Adolescent/Young Adult Hematopoietic Stem Cell Transplant Recipients. Diabetes Technol Ther. 2023 Feb;25(2):116-121. doi: 10.1089/dia.2022.0246. Epub 2022 Dec 29. PMID 36511871
- [Derived] Sopfe J, Pyle L, Keating AK, Campbell K, Liu AK, Wadwa RP, Verneris MR, Giller RH, Forlenza GP. Malglycemia is associated with poor outcomes in pediatric and adolescent hematopoietic stem cell transplant patients. Blood Adv. 2019 Feb 12;3(3):350-359. doi: 10.1182/bloodadvances.2018021014. PMID 30718242